CLINICAL TRIAL: NCT06911840
Title: Assessment of Male Factor Infertility Across India: An Observational Cross-Sectional Study Using the Aphrodite Criteria, a Hospital-based Study
Brief Title: Male Factor Infertility Across India Using Aphrodite Criteria
Acronym: APHR
Status: Not yet recruiting | Type: Observational
Sponsor: Indira IVF Hospital Pvt Ltd (Other)
Responsible Party: Principal Investigator, Dr Vipin Chandra, Chief Clinical Lab Operations, Indira IVF Hospital Pvt Ltd
Other Study IDs: IIHL/UDR/P/02_2024
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Male Infertility Due to Azoospermia
Keywords: Male infertility; Azoospermia; Aphrodite criteria; Prevelance
MeSH Terms: conditions — Infertility, Male; Azoospermia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All the male population visiting IVF centre
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
Study Purpose:

The purpose of this study is to conduct an observational cross-sectional analysis of male factor infertility across diverse regions of India utilizing the Aphrodite Criteria. This novel patient classification system offers a systematic approach to describing and managing male infertility, particularly for hypogonadal males with idiopathic infertility. The study aims to evaluate the current state of male fertility across India and identify any regional variations in male reproductive health and hypogonadism, which may be influenced by environmental, lifestyle, and genetic factors.

Study Objective:

The primary objective of this study is to conduct an observational cross-sectional analysis of male factor infertility across various regions of India using the Aphrodite Criteria. To reveal the prevalence and determinants of male factor infertility across different regions of India.

Hypothesis:

We hypothesize that there are significant regional differences in male factor infertility characteristics across India, with variations in sperm quality and testicular function due to diverse environmental, lifestyle, and genetic factors. Additionally, we hypothesize that the application of the Aphrodite Criteria will provide a more detailed classification of male infertility compared to conventional semen analysis and that certain lifestyle factors such as smoking, obesity, and occupational exposures will be associated with poorer sperm quality and testicular function.

Study Population:

The study population will consist of male patients visiting clinics across different IVF centers in India. The total sample size includes subjects from five groups with the following distribution:

35 subjects in Group I ; 416 subjects in Group II; 270 subjects in Group III; 152 subjects in Group IV; 216 subjects in Group V

The total sample size for all groups will be 1,090 subjects.

ELIGIBILITY:
Inclusion Criteria:

* All male visiting IVF clinic willingly giving consent for andrological evaluation.

Exclusion Criteria:

* NONE

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male attending IVF Clinic
Study Population: All male visiting IVF clinics across different centres
Sampling Method: Non-Probability Sample
Enrollment: 1090 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Prevalence of male infertility across the country | 6 months
  Overall prevalence of male infertility according to the Aphrodite criteria in India.

SECONDARY OUTCOMES:
Prevalence of male infertility across various geographical distribution | 6 months
  Prevalence of male infertility according to the Aphrodite criteria in different regions of India.
Factors associated with male infertility | 6 months
  Factors associated with male infertility according to the Aphrodite criteria, both overall and stratified by region

CONTACTS AND LOCATIONS:
Locations (1):
- Indira IVF Hospital, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Yes
The following supporting information will be made available as part of the data sharing plan:
  Study Protocol
  Available upon request or publication of study results.
  Statistical Analysis Plan (SAP)
  Will be shared with interested parties upon completion of the study.
  Informed Consent Form (ICF)
  A copy of the ICF will be available upon request from participating sites.
  Clinical Study Report (CSR)
  The final CSR will be shared once the study results are finalized and published.
  Analytic Code
  Will be shared alongside the study results for transparency and reproducibility of the findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study and on request
Access Criteria: Academic researchers, clinicians, and scientists involved in related fields of study.
  Regulatory Bodies: Organizations such as ethics committees, health authorities, and regulatory agencies that require access for monitoring and compliance purposes.
  Collaborators and Partners: Institutions or organizations collaborating on the study, subject to agreements for data sharing and confidentiality.
  What They Will Be Able to Access:
  Study Protocol: Complete details regarding the study design, objectives, and methodology.
  Statistical Analysis Plan (SAP): Full plan for data analysis, statistical methods, and handling of results.
  Informed Consent Form (ICF): Document outlining the consent process and participant rights, shared with participating researchers and ethics boards.
  Clinical Study Report (CSR): The final comprehensive report including all study findings, results, and conclusions.
  Analytic Code: The code used for statistical analysis, available for validation and reproducibility

REFERENCES:
- [Result] Esteves SC, Yarali H, Vuong LN, Carvalho JF, Ozbek IY, Polat M, Le HL, Pham TD, Ho TM. Low Prognosis by the POSEIDON Criteria in Women Undergoing Assisted Reproductive Technology: A Multicenter and Multinational Prevalence Study of Over 13,000 Patients. Front Endocrinol (Lausanne). 2021 Mar 12;12:630550. doi: 10.3389/fendo.2021.630550. eCollection 2021. PMID 33790862
- [Result] May WL, Johnson WD. A SAS macro for constructing simultaneous confidence intervals for multinomial proportions. Comput Methods Programs Biomed. 1997 Jul;53(3):153-62. doi: 10.1016/s0169-2607(97)01809-9. PMID 9230450
- [Result] Esteves SC, Humaidan P, Ubaldi FM, Alviggi C, Antonio L, Barratt CLR, Behre HM, Jorgensen N, Pacey AA, Simoni M, Santi D. APHRODITE criteria: addressing male patients with hypogonadism and/or infertility owing to altered idiopathic testicular function. Reprod Biomed Online. 2024 Apr;48(4):103647. doi: 10.1016/j.rbmo.2023.103647. Epub 2023 Oct 29. PMID 38367592